CLINICAL TRIAL: NCT00953901
Title: Restrictive Versus Liberal Fresh Frozen Plasma Transfusion Prior to Low-Risk Invasive Procedures in Hospitalized Patients.
Brief Title: Is Plasma Transfusion Beneficial Prior to Low-Risk Procedures in Hospitalized Patients With Blood Clotting Abnormalities?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2247-05
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Blood Coagulation, Disorders; Surgical Procedures, Minimally Invasive
MeSH Terms: conditions — Hemostatic Disorders

INTERVENTIONS:
Drug: Fresh Frozen Plasma Transfusion

SUMMARY:
Blood clotting abnormalities or problems that happen during surgery ? even minor surgery ? are serious because of the possibility of serious bleeding that cannot be stopped. The current standard practice for people with clotting abnormalities is to transfuse additional blood before the surgery, in an effort to decrease bleeding problems. However, transfusing blood before the surgery is not very effective in decreasing bleeding complications. In addition, it may be associated with other complications, including fluid buildup and swelling in the lungs. For this study, a person with a mild clotting problem is defined as one with an INR (International Normalized Ratio) between 1.5 and 3. Severe clotting is defined as an INR greater than 3. This study will aim to test if limiting or restricting transfusion for those patients with severe clotting problems (an INR greater than 3) will result in fewer transfusion problems and fewer unnecessary transfusions in comparison with the current, more liberal, transfusion use for all patients with both mild and severe clotting problems (an INR greater than 1.5).The investigators will also determine if liberal blood transfusion decreases the risk of bleeding after surgical procedures.

DETAILED DESCRIPTION:
While the restrictive red cell transfusion practice has become a standard of care in the acutely ill, data on the use of fresh frozen plasma (FFP) are limited. FFP transfusion may not only be poorly effective in prevention of bleeding complications but is associated with significant complications. In a retrospective cohort of critically ill non-surgical patients with abnormal international normalized ratio (INR), we have observed significant variability in the practice of FFP transfusion. Rather than a benefit with liberal use, more adverse effects were observed, in particular pulmonary edema and acute lung injury. Our overall goal is to improve the safety of blood product transfusion and prevent pulmonary complications. Here we propose a randomized clinical trial of restrictive (INR 1.6-3) versus liberal (FFP transfusion to keep INR < 1.6) FFP transfusion prior to commonly performed invasive procedures (thoracocentesis, abdominal paracentesis and central venous cannulation). We will use the following outcome measures to compare the differences between the two groups: 1. New onset pulmonary edema; 2. Postprocedural bleeding complications; 3. Number of blood product transfusions; 4. Hospital mortality and 5. Length of intensive care unit and hospital stay. The results of this study will form the basis for future multicenter clinical trials with implications for worldwide transfusion practice.

ELIGIBILITY:
Inclusion:

* Consenting hospitalized adult
* (>18 years)
* Patients with abnormal INR (INR 1.6-3) due to either vitamin K depletion or antagonism (Coumadin and/or broad spectrum antibiotics) or liver insufficiency
* Patients who are about to undergo one of the three common minimally invasive procedures (thoracocentesis, abdominal paracentesis, and central vein cannulation)

Exclusion:

* None

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-07; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
New onset pulmonary edema

SECONDARY OUTCOMES:
Postprocedural bleeding complications
Number of blood product transfusions
Hospital mortality
Length of intensive care unit and hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States